CLINICAL TRIAL: NCT05644717
Title: Effects of Ertugliflozin on Liver Fat, Liver Fibrosis & Glycemic Control in Subjects With Type 2 Diabetes Mellitus (T2DM) & Non-Alcoholic Fatty Liver Disease /Non-Alcoholic Steatohepatitis
Brief Title: Effect of Erugliflozin On Liver Fat, Liver Fibrosis and Glycemic Control in Type II DM Patients With NASH/NAFLD
Acronym: Ertu-NASH
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Getz Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GTZ_DM_007_22
Record Dates: First submitted 2022-11-18; First posted 2022-12-09 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Liver Fat; Liver Fibrosis; Glycemic Control; Body Weight Changes; Waist Circumference; Tolerance
MeSH Terms: conditions — Fatty Liver; Liver Cirrhosis; Body Weight Changes | interventions — ertugliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ertugliflozin (Experimental): Ertugliflozin 5/15mg once daily with standard of care
  Interventions: Drug: Ertugliflozin 5 mg, 15mg

INTERVENTIONS:
Drug: Ertugliflozin 5 mg, 15mg — Ertugliflozin 5/15mg once daily in addition to standard of care

SUMMARY:
Open-label, prospective, single-arm, multicenter study to determine effects of Ertugliflozin on liver fat, liver fibrosis & glycemic control in subjects with Type 2 Diabetes Mellitus (T2DM) with Non-Alcoholic Fatty Liver Disease (NAFLD)/Non-Alcoholic Steatohepatitis (NASH)

ELIGIBILITY:
Inclusion Criteria:

* Patient able to provide written informed consent
* Adult males & females between 18 to 65 years
* SGLT2i and insulin naïve patients
* BMI >23 Kg/m2
* HbA1C % ≥ 6.5 to 10
* Documented hepatic steatosis or fatty liver disease on Ultrasound
* Patient with Type II Diabetes Mellitus

Exclusion Criteria:

* History of use of SGLT 2 inhibitors or Glucagon-like peptide (GLP) 1 agonist or insulin; 3 months prior to enrollment in the study.
* Pioglitazone use in the past 6 months
* History of vitamin E use (400mg twice daily) 3 months prior to enrollment in the study.
* History of anti-obesity medication or weight loss procedure (bariatric surgery) use within 3 months prior to enrollment in the study.
* History of uncontrolled Endocrine disorder (for example uncontrolled hypothyroidism, or that requires frequent dose adjustment, or Cushing's syndrome)
* History of liver disease including viral hepatitis, auto-immune hepatitis, liver cirrhosis, hepatocellular carcinoma and/or HIV
* History of recurrent UTIs and mycotic infection.
* Severely ill patients (who have high grade fever, sepsis or acute infection)
* Pregnant woman, lactating woman or planning pregnancy during study duration
* History of Drug-induced liver disease (e.g. amiodarone, valproate, tamoxifen, methotrexate, steroids (including homeopathic medicines).
* History of active substance abuse (cannabinoid-derived substances like heroin, cocaine, amphetamines) based on history and/or laboratory tests
* Alcohol intake 10 - 30 g/day (three drinks per day) within the previous year
* Active substance abuse such as acetaminophen over-use, hashish, tobacco products, heroin, cocaine or amphetamines.
* Severe hepatic impairment ( AST & ALT levels > 3 times upper limit normal

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Radiologic liver parameters | up to 24 weeks
  Number of participants reported change in liver fat content from baseline, as quantified by fibroscan

SECONDARY OUTCOMES:
HbA1c% levels compare with baseline in 6 months | up to 24 weeks
  Efficacy
Change in body weight compare with baseline in 6 months | up to 24 weeks
  Body Weight
Change in waist circumference compare with baseline in 6 months | up to 24 weeks
  Waist Circumference
Fibrosis 4 score levels compare with baseline in 6 months | up to 24 weeks
  Fibrosis Scoring < 1.45 indicates Fibrosis Stage 0-2, 1.45 to 3.25 is deemed indeterminate fibrosis stage, > 3.25 indicates Fibrosis stage 3-4
Non-Alchoholic Fatty Liver Disease Fibrosis Score levels compare with baseline in 6 months | up to 24 weeks
  Non-Alchoholic Fatty Liver Disease Fibrosis Scoring, < -1.455 indicates Fibrosis Stage 0-2,
  -1.455 to 0.676 is considered indeterminate fibrosis stage, > 0.676 indicates Fibrosis Stage 3-4
Frequency of adverse events in 6 months | up to 24 weeks
  Safety

CONTACTS AND LOCATIONS:
Overall Officials: Umar Raja, MBBS, Principal Investigator — Shifa International Hospital
Locations (1):
- North west general hospital, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hu M, Phan F, Bourron O, Ferre P, Foufelle F. Steatosis and NASH in type 2 diabetes. Biochimie. 2017 Dec;143:37-41. doi: 10.1016/j.biochi.2017.10.019. Epub 2017 Oct 31. PMID 29097281
- [Background] Targher G, Byrne CD, Lonardo A, Zoppini G, Barbui C. Non-alcoholic fatty liver disease and risk of incident cardiovascular disease: A meta-analysis. J Hepatol. 2016 Sep;65(3):589-600. doi: 10.1016/j.jhep.2016.05.013. Epub 2016 May 17. PMID 27212244
- [Background] Mantovani A, Byrne CD, Bonora E, Targher G. Nonalcoholic Fatty Liver Disease and Risk of Incident Type 2 Diabetes: A Meta-analysis. Diabetes Care. 2018 Feb;41(2):372-382. doi: 10.2337/dc17-1902. PMID 29358469
- [Background] Mantovani A, Zaza G, Byrne CD, Lonardo A, Zoppini G, Bonora E, Targher G. Nonalcoholic fatty liver disease increases risk of incident chronic kidney disease: A systematic review and meta-analysis. Metabolism. 2018 Feb;79:64-76. doi: 10.1016/j.metabol.2017.11.003. Epub 2017 Nov 11. PMID 29137912
- [Background] Schuppan D, Schattenberg JM. Non-alcoholic steatohepatitis: pathogenesis and novel therapeutic approaches. J Gastroenterol Hepatol. 2013 Aug;28 Suppl 1:68-76. doi: 10.1111/jgh.12212. PMID 23855299
- [Background] Gusdon AM, Song KX, Qu S. Nonalcoholic Fatty liver disease: pathogenesis and therapeutics from a mitochondria-centric perspective. Oxid Med Cell Longev. 2014;2014:637027. doi: 10.1155/2014/637027. Epub 2014 Oct 13. PMID 25371775